CLINICAL TRIAL: NCT04688645
Title: Treatment With Balanced Crystalloid Solutions in the Early Phase of Acute Pancreatitis
Brief Title: Balanced Crystalloid Solutions for Acute Pancreatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Rijeka (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Principal Investigator, Goran Poropat, Asst. Prof., University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: uniri-biomed-18-154
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Plasmalyte A; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balanced crystalloid solution (Experimental): Balanced crystalloid solution - Plasmalyte.
  Interventions: Drug: Balanced crystalloid solution
- Normal saline (Active Comparator): 0.9% sodium chloride solution.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Balanced crystalloid solution — Balanced crystalloid solution (Plasmalyte) given as an initial bolus of 10 ml/kg body weight within the first 60 min after randomization, and then continued at a rate of 2 ml/kg body weight during the next 72 hours. If needed boluses may be repeated.
  Other Names: Plasmalyte; balanced crystalloids
  Arms: Balanced crystalloid solution
Drug: Normal saline — 0.9% sodium chloride solution given as an initial bolus of 10 ml/kg body weight within the first 60 min after randomization, and then continued at a rate of 2 ml/kg body weight during the next 72 hours. If needed boluses may be repeated.
  Other Names: Saline; 0.9% sodium chloride solution
  Arms: Normal saline

SUMMARY:
Patients diagnosed with acute pancreatitis regardless of etiology, severity of disease, and prior attacks will be randomized in two groups. The intervention group will receive a balanced crystalloid (Plasmalyte) at a rate of 10 ml/kg during the first 60 min and then continued at 3 ml/kg/h for the next 72 hours. The control group will receive normal saline at the same rate.

ELIGIBILITY:
Inclusion Criteria:

- patients diagnosed with acute pancreatitis based on the revised Atlanta criteria who present to our hospital within 48 hours of symptoms onset, regardless of etiology, severity of disease, or prior episodes of acute pancreatitis

Exclusion Criteria:

* chronic pancreatitis
* liver cirrhosis (Child-Pugh B and C)
* chronic hearth failure (NYHA>II)
* acute coronary syndrome
* cardiovascular intervention within 60 days before randomization
* chronic obstructive pulmonary disease dependent of home oxygenator or acute exacerbation of chronic obstructive pulmonary disease
* chronic kidney disease (eGFR <30 ml/min/1.73 m2)
* concomitant biliary infection (cholecystitis, cholangitis)
* severe autoimmune disease
* chronic active infection (TBC, AIDS)
* metastatic malignant disease
* primary pancreatic neoplasm
* patients transferred from other hospitals
* pregnancy and ongoing breastfeeding
* not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with New Onset Systemic inflammatory response syndrome (SIRS) | 30 days
  Body temperature less than 36 °C (96.8 °F) or greater than 38 °C (100.4 °F); heart rate greater than 90 beats per minute; tachypnea (high respiratory rate), with greater than 20 breaths per minute or, an arterial partial pressure of carbon dioxide less than 4.3 kilopascals (32 mmHg); white blood cell count less than 4000 cells/mm³ (4 x 109 cells/L) or greater than 12,000 cells/mm³ (12 x 109 cells/L) or the presence of greater than 10% immature neutrophils.

SECONDARY OUTCOMES:
Mortality | 30 days
  Number of death cases
Number of participants with organ failure (transitory and persistent) | 30 days
  Organ failure defined according to the modified Marshall criteria
Number of participants with local complications | 30 days
  Local complications including:
  * acute peripancreatic fluid collection
  * acute necrotic collection
  * pseudocyst
  * walled-off necrosis
Number od participants with systemic complications | 30 days
  Worsening of existing concomitant diseases
Number of participants with infected pancreatic necrosis | 30 days
  Defined by positive cultures from fine-needle aspiration of necrotic tissue or by the combination of clinical deterioration with clinical signs of infection and presence of gas within the necrotic tissue on imaging in cases of culture-negative, but highly suspicious cases.
Number of participants needing endoscopic / percutaneous / surgical interventions | 30 days
  In cases when presence of local infection or local complications (i.e. collection compressing surrounding organs and causing symptoms) requires an intervention
Length of hospital stay | 30 days
  Number of days in hospital, from admission to discharge or death.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No